CLINICAL TRIAL: NCT02807337
Title: Supersaturated Calcium Phosphate Oral Rinse (Caphosol®) For the Prevention of Oral Mucositis in Children Undergoing Chemotherapeutic Treatments
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R16021
Record Dates: First submitted 2016-06-07; First posted 2016-06-21 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-01

CONDITIONS: Cancer
Keywords: Oral mucositis
MeSH Terms: conditions — Neoplasms; Stomatitis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Caphosol rinse group (Experimental): Caphosol consists of two solutions (A and B) which are mixed immediately before use. Caphosol mouth rinse will begin concomitantly (the same day) with the beginning of chemotherapeutic drugs. It will be continued for seven consecutive days.
  Interventions: Drug: Caphosol
- 0,9% NaCl group. (Active Comparator): 0,9% NaCl consists of two solutions (A and B). Two vials of 0.9% NaCl will be mixed to maintain blinding. The study mouth rinse will begin concomitantly (the same day) with the beginning of chemotherapeutic drugs. It will be continued for seven consecutive days.
  Interventions: Drug: 0,9% NaCl

INTERVENTIONS:
Drug: Caphosol
  Arms: Caphosol rinse group
Drug: 0,9% NaCl
  Arms: 0,9% NaCl group.

SUMMARY:
Prospective double-blinded randomized clinical study. Aim of the study is to compare the effectiveness of Caphosol mouth rinses in prevention of oral mucositis as compared to 0.9% NaCl rinses. Patients will be randomized to receive either Caphosol or 0.9% NaCl rinses four times a day for seven days from the beginning of chemotherapeutic regimen. The same patient will be given the opposite rinse during the next chemotherapeutic regimen, so everyone will get both mouth rinses once during the trial.

DETAILED DESCRIPTION:
The study will be a double-blinded study so that the researchers or research nurses and the patients/parents are unaware of the solution used (Caphosol vs 0.9% NaCl). They both taste very similar and are packaged to ampules similar to each other. Since Caphosol consists of two solutions (A and B) which are mixed immediately before use, the investigators will apply the same procedure also in case of 0.9% NaCl solution (two vials of 0.9% NaCl will be mixed) to maintain blinding. Caphosol and 0.9% NaCl rinses will be relabeled to maintain blinding. Every patient will participate two times in the study. The treatment group allocation is based on randomization and will be performed once before participation for the first time. During another chemotherapeutic regimen, the same patient will automatically use another mouth rinse (Group 1 => Group 2 and Group 2 => Group 1). This dependence-effect caused by observations gathered from same patients will be taken into account when analysing the data. Blinding will be maintained throughout the study.

The investigators estimate that occurrence of oral mucositis as a side effect of chemotherapeutic treatment differs by 3-fold in different study arms (10% in Caphosol group, and 30% in 0.9% NaCl group). Power calculations using power of 0.8 and p-value of 0.05 indicate that the 70 children are needed to be recruited into each arm, i.e. two repeated measurements from 70 children are needed to have adequate statistical power. A drop-out of approximately 3-5% of patients has been taken into account and therefore the investigators plan to recruit 75 patients. Randomization will be performed using freely available and web-based MINIM-randomization software.

The data analysis will be performed on intention-to-treat principle. Mixed-effect regression methods will be used due to repeated observation within study subjects.

Specific methods used for this study:

* Oral mucositis will be assessed daily for all patients at the oncology ward and at home by use of the Children International Mucositis Evaluation Scale and World Health Organization oral mucositis scale.
* In the beginning of study, initial clinical evaluation will be performed by a pediatric dentist. During the stay at hospital, parents/patients (or nurses) will fill in the oral mucositis scales. At home, the patients/parents fill the scales. Scales will be filled in once a day for 14 consecutive days. Caphosol / 0.9% NaCl rinse treatment will last for only 7 consecutive days.
* The available medical and dental records will be audited for the frequency of oral mucositis.
* Oral samples will be collected by a pediatric dentist, and bacterial analyses will be performed by microbiologist at University of Tampere.
* Laboratory values and pain medications will be retrieved from electronic patient files (MIRANDA/Fimlab).
* Blood tests will be collected for possible later use in genetic studies.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric cancer patients aged 2 - 17.99 years old
2. Patients diagnosed with solid or hematological malignancy and receiving chemotherapeutic drugs.
3. Use of the following mucosa-breaking chemotherapeutic drugs: high-dose methotrexate, any anthracycline (doxorubicin, daunorubicin, idarubicin, mitoxantrone), and cisplatin.
4. Protocol must include potential mucosa-breaking chemotherapeutic cycles at least twice in the protocol.

Exclusion Criteria:

1. Patients younger than 2 years old or older than 18 years.
2. Patients who have mucositis at the start of chemotherapeutic regimen.
3. Less than three weeks from previous treatment ("washout" period).
4. High-dose chemotherapy with stem cell transplantation patients.
5. Induction treatment (leukemia).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Oral mucositis will be assessed daily for all 75 pediatric patients at the oncology ward and at home by use of the Children International Mucositis Evaluation Scale (ChIMES scale) and WHO oral mucositis scale. | 3 years
  ChIMES Scale - illustrations of faces with expressions corresponding to the following scores:children will select the face that best describes how they are feeling. Oral samples will be collected by a pediatric dentist, and bacterial analyses will be performed later on. Also, blood tests will be collected for possible later use in genetic studies.

CONTACTS AND LOCATIONS:
Overall Officials: Egle Immonen, Principal Investigator — Tampere University Hospital
Locations (3):
- Finland (3):
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Immonen E, Paulamaki L, Piippo H, Nikkila A, Aine L, Peltomaki T, Lohi O, Parikka M. Oral microbiome diversity and composition before and after chemotherapy treatment in pediatric oncology patients. BMC Oral Health. 2025 Jul 2;25(1):981. doi: 10.1186/s12903-025-06405-4. PMID 40604730
- [Derived] Immonen E, Aine L, Nikkila A, Parikka M, Gronroos M, Vepsalainen K, Palmu S, Helminen M, Peltomaki T, Lohi O. Randomized controlled and double-blinded study of Caphosol versus saline oral rinses in pediatric patients with cancer. Pediatr Blood Cancer. 2020 Oct;67(10):e28520. doi: 10.1002/pbc.28520. Epub 2020 Jul 29. PMID 32725875